CLINICAL TRIAL: NCT02754427
Title: Pilot Study for a Prospective Surveillance Program for Rehabilitation Following Surgery for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H12-01773
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: Surveillance; Physiotherapy; Arm morbidity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective Surveillance Group (Experimental): Women assigned to surveillance group were assessed for arm morbidity at pre-surgery and at 3, 6, and 9 months post-surgery. If arm morbidity was detected at any time-point post-surgery, then a physiotherapy intervention was prescribed.
  Interventions: Behavioral: Prospective Surveillance Group
- Education Group (Active Comparator): Participants in the education group received the usual post-operative follow-up.
  Interventions: Behavioral: Education Group

INTERVENTIONS:
Behavioral: Prospective Surveillance Group — Participants received a pre-surgery arm assessment for shoulder mobility, upper body muscle strength, upper body function, and arm volume. Same assessment was repeated at 12 months post-surgery. After surgery, participants randomized to the surveillance group underwent the same arm assessment at 3, 6, and 9 months post-surgery. If arm morbidity was detected at any of those time points, then the participant was referred to individual physiotherapy treatment until the issue was resolved.
  Other Names: Prospective surveillance for arm morbidity and physiotherapy treatment
  Arms: Prospective Surveillance Group
Behavioral: Education Group — Participants received a pre-surgery arm assessment for shoulder mobility, upper body muscle strength, upper body function, and arm volume. Same assessment was repeated at 12 months post-surgery. After surgery, participants randomized to the education group were asked to attend three patient education sessions on nutrition, stress management, and fatigue management of approximately 1 hour, delivered at 3, 6, and 9 months by study staff.
  Other Names: Attention Control Group
  Arms: Education Group

SUMMARY:
Breast cancer treatment often results in long-term arm morbidity. A prospective surveillance model with arm assessment pre-surgery followed by ongoing surveillance and targeted physiotherapy treatment after breast cancer surgery may improve early detection and management of arm morbidity. This study aims to determine the effect of prospective surveillance to target physiotherapy on the prevalence of arm morbidity in the surveillance group compared to control group at 12-months after breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 30-75 years; receiving surgery for breast cancer, including those who will have immediate breast reconstruction.

Exclusion Criteria:

* prior breast cancer surgery; a pre-existing shoulder pathology on the side of breast surgery that limits shoulder range of motion <75% of non-affected side; or a diagnosis of primary lymphedema

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Campbell, PhD, Principal Investigator — kristin.campbell@ubc.ca

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Surveillance Group | Education Group
Started | 21 | 20
Completed | 21 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective Surveillance Group | Education Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.05 (6.4) | 53.25 (10.0) | 54.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0
  Ethnicity: Not Hispanic or Latino | 21 | 20 | 41
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Arm Morbidity at 12 Months Post-surgery - Shoulder Mobility
Description: Arm morbidity due to decreased shoulder mobility was defined as ≥10% decrease in mobility from pre-surgery. This was measured using a goniometer and evaluated the degrees of shoulder mobility in flexion, abduction and external rotation.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Surveillance Group | Education Group
Number analyzed (Participants) | 21 | 19
Participants | 5 | 7

2. Primary Outcome: Number of Participants With Arm Morbidity at 12 Months Post-surgery - Upper Body Muscle Strength
Description: Arm morbidity due to decreased upper body muscle strength was defined as ≥25% decrease in muscle strength from pre-surgery. This was measured using a hand-held dynamometer and evaluated in kilograms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Surveillance Group | Education Group
Number analyzed (Participants) | 21 | 19
Participants | 1 | 4

3. Primary Outcome: Number of Participants With Arm Morbidity at 12 Months Post-surgery - Upper Body Function
Description: Arm morbidity due to decreased upper body function was defined as ≥10 points decrease in function from pre-surgery. This was measured using the Upper Extremity Functional Index that scores 0 to 80, with higher scores indicating greater level of function.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Surveillance Group | Education Group
Number analyzed (Participants) | 21 | 19
Participants | 5 | 3

4. Primary Outcome: Number of Participants With Arm Morbidity at 12 Months Post-surgery - Arm Volume
Description: Arm morbidity due to increase in arm volume was defined as a ≥200 mL increase from pre-surgery. Arm volume was measured using a perometer.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Surveillance Group | Education Group
Number analyzed (Participants) | 21 | 19
Participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Prospective Surveillance Group | Education Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No